CLINICAL TRIAL: NCT02542878
Title: Acute Effects of Foam Rolling Self-application on Isometric Back Extension Endurance on Basketball Players. A Pilot Study.
Brief Title: Effect of Myofascial Release by Foam Rolling on Back Muscles Endurance
Acronym: FR-Lumbar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Sergio Hernandez Sanchez, Physical Therapist (PT), Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DPC-SHS-01.15
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Back Injuries
Keywords: myofascial release; back extensors endurance; foam roller; sport
MeSH Terms: conditions — Back Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOAM ROLLER (Experimental): Treatment with foam roller will be applied for 60 seconds to this group. Subjetc lye in supine position over the foam roller placed on back muscle extensors. Then, they must slide the body on the device, from postero-superior iliac spine to the dorsal zone.
  A brief explanation of this self-application will be showed prior the intervention.
  Interventions: Device: Foam roller
- PLACEBO (Placebo Comparator): An intervention similar (position and time) to the experimental group will be done, but the used device will be a very soft roller not compressing the contact zone.

INTERVENTIONS:
Device: Foam roller — A bout of 60 seconds of myofascial release with foam roller
  Arms: FOAM ROLLER

SUMMARY:
This study evaluate the effect of the a low back self-application of myofascial release using a foam rolling on back muscles endurance measured by the Biering-Sorensen test.

DETAILED DESCRIPTION:
Self-myofascial release performed with a foam roller is an incoming technique what is very popular in sport. Scientific literature currently suggests that the effects of self-myofascial release are mediated by the stimulation over neural and connective tissue. There is evidence that this stimulation could improve the maximum range of motion and decrease muscle soreness. Nonetheless, there is few evidence about the effects of self-myofascial release on muscle endurance.

Given the increased use of autonomously (self-treatment) in the athlete population, this study aims to assess the effect of a low back short application (60 seconds) on the back extensor muscles endurance measured by the Biering-Sorensen test.

With the obtained results we want to elaborate an evideced based recommendation about its use prior to physical activity or sports competition.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players, between 18-25 years who participate on a official league and do regular physical training (4 training sessions 1.5 hours each and a competitive session a week)
* Be able to read and understand the premises of the informed consent of the study.

Exclusion Criteria:

* to present some osteo-articular and / or muscle-tendon pathology that could be exacerbated by the implementation of the Biering-Sorensen test or by the intervention with foam compression.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Isometric back extensors endurance | 1 day
  Biering-Sorensen test will be applied, which consists is to keep the trunk straight and parallel to the floor as long as possible, with lower limb fixed to the table up to the antero-superior iliac spine in prone position.

CONTACTS AND LOCATIONS:
Overall Officials: SERGIO HERNANDEZ-SANCHEZ, PT PhD Stud, Principal Investigator — Professor Physiotherapy Degree

REFERENCES:
- [Background] Mohr AR, Long BC, Goad CL. Effect of foam rolling and static stretching on passive hip-flexion range of motion. J Sport Rehabil. 2014 Nov;23(4):296-9. doi: 10.1123/jsr.2013-0025. Epub 2014 Jan 21. PMID 24458506
- [Background] Macdonald GZ, Button DC, Drinkwater EJ, Behm DG. Foam rolling as a recovery tool after an intense bout of physical activity. Med Sci Sports Exerc. 2014 Jan;46(1):131-42. doi: 10.1249/MSS.0b013e3182a123db. PMID 24343353
- [Background] Sullivan KM, Silvey DB, Button DC, Behm DG. Roller-massager application to the hamstrings increases sit-and-reach range of motion within five to ten seconds without performance impairments. Int J Sports Phys Ther. 2013 Jun;8(3):228-36. PMID 23772339
- [Background] MacDonald GZ, Penney MD, Mullaley ME, Cuconato AL, Drake CD, Behm DG, Button DC. An acute bout of self-myofascial release increases range of motion without a subsequent decrease in muscle activation or force. J Strength Cond Res. 2013 Mar;27(3):812-21. doi: 10.1519/JSC.0b013e31825c2bc1. PMID 22580977
- [Background] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488
- [Background] Halperin I, Aboodarda SJ, Button DC, Andersen LL, Behm DG. Roller massager improves range of motion of plantar flexor muscles without subsequent decreases in force parameters. Int J Sports Phys Ther. 2014 Feb;9(1):92-102. PMID 24567860
- [Background] Coorevits P, Danneels L, Cambier D, Ramon H, Vanderstraeten G. Assessment of the validity of the Biering-Sorensen test for measuring back muscle fatigue based on EMG median frequency characteristics of back and hip muscles. J Electromyogr Kinesiol. 2008 Dec;18(6):997-1005. doi: 10.1016/j.jelekin.2007.10.012. Epub 2008 Apr 8. PMID 18396410
- [Background] Evans K, Refshauge KM, Adams R. Trunk muscle endurance tests: reliability, and gender differences in athletes. J Sci Med Sport. 2007 Dec;10(6):447-55. doi: 10.1016/j.jsams.2006.09.003. Epub 2006 Dec 1. PMID 17141568
- [Background] Demoulin C, Vanderthommen M, Duysens C, Crielaard JM. Spinal muscle evaluation using the Sorensen test: a critical appraisal of the literature. Joint Bone Spine. 2006 Jan;73(1):43-50. doi: 10.1016/j.jbspin.2004.08.002. PMID 16461206
- [Background] Suter E, Lindsay D. Back muscle fatigability is associated with knee extensor inhibition in subjects with low back pain. Spine (Phila Pa 1976). 2001 Aug 15;26(16):E361-6. doi: 10.1097/00007632-200108150-00013. PMID 11493865